CLINICAL TRIAL: NCT05302440
Title: The Perceived Efficiency and Acceptability of Remote Real-time Health Monitoring System in Elderly Residential Setting and Community Isolation Facility
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: Haven of Hope Hospital (Other); The Social Innovation and Entrepreneurship Development Fund, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Derek Yee-Tak Cheung, Assistant Professor, The University of Hong Kong
Other Study IDs: HKU_real-time_monitor_v3
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Results first posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-01

CONDITIONS: Technology
Keywords: Gerontechnology; Smart Healthcare Device; Digital Health Technology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- single-group: All care staff who manage the system will complete a very brief survey (1-minute) after each work shift for 14 days. Detection of abnormal vital signs will be recorded by the system. Hospital admission and further medical assistance due to the use of the system will be documented by the care team. The staff will be interviewed about their perceived benefits and acceptability of the system.
  Interventions: Device: remote real-time health monitoring system with ring-like sensor

INTERVENTIONS:
Device: remote real-time health monitoring system with ring-like sensor — The remote monitoring system will constantly record the temperature, pulse and SpO2 of the residents wearing the equipment. When the staff find abnormal vital signs, they will provide further medical assistance. All care staff who manage the system will be complete a very brief survey (1-minute) after each work shift for 14 days.

SUMMARY:
The study has 3 primary research questions and 6 secondary research questions targeting care staff in the setting of residential care homes for the elderly. The 3 primary research questions are:

1. Will care staff perceive the remote real-time health monitoring system with ring-like sensor as efficient?
2. Will the system facilitate any early detection of abnormal vital signs?
3. Will the system facilitate early delivery of medical support?

   The 6 secondary research questions are:
4. What are the numbers of hospital admissions and further medical assistance due to the adoption of the system?
5. Will the system reduce the stress level of the care staff?
6. What are the perceived benefits and acceptability of the care staff towards the system?
7. What should be considered when developing the evaluation framework for the adaption of the system in elderly residential setting?
8. Are there any barriers and difficulties in the set-up of the system?
9. What are the concerns in choosing wireless or cable connection for the monitoring device?

DETAILED DESCRIPTION:
Study design

This is a single-group 4-week trial of using the remote health monitoring system. All care staff who manage the system will complete a very brief survey (1-minute) after each work shift for 2 weeks. Detection of abnormal vital signs will be recorded by the system. Hospital admission and further medical assistance due to the adoption of the system will be documented by the care team. The care staff will be interviewed about their perceived benefits and acceptability of the system.

Subjects

Care staff in Haven of Hope Woo Ping Care & Attention Home and Haven of Hope Nursing Home who are responsible to set up and operate real-time remote health monitoring system will be recruited. They also need to be able to read and understand Chinese.

Procedures

Implementation

The remote monitoring system will record the temperature, pulse and oxygen saturation (SpO2) of the residents wearing the equipment every minute. When the staff find abnormal vital signs, they will provide further medical assistance. After every shift during the trial period for 2 weeks, they will fill in a 1-minute survey.

Data collection

The remote monitoring system will remotely and real-time record the temperature, pulse and SpO2 of the residents wearing the sensor. The sensor is like a ring that wraps a finger. When the staff are notified of any abnormal vital signs by the system via screen display and notification sound, they will deliver further medical assistance. Hospital admission and further medical assistance due to the adoption of the system will be documented by the care team under pre-existing practice. After every shift during the trial period for 2 weeks, the staff will fill in a 1-minute survey about their operation and perceived efficiency of the system, such as facilitating more frequent monitoring of particular residents' vital signs, the provision of further medical assistance, perceived time saving in monitoring vital signs, and acceptability of the system. They could record their experience of using the system in a messaging mobile phone app in audio format. If they fill in the survey for fewer than 10 times during the 2 weeks, they would be invited to continue to fill in the survey after work shift after the 2 weeks until they fill in it for at least 10 times. Meanwhile, as a staff may complete more than 1 shift per day, they would not be invited to fill in the survey after having completed it for 12 items. All data collected that is related to residents is not identifiable.

There are two parts of the qualitative sub-study. When the system is set up, the unit in-charge and care staff responsible to set up the system from each participating unit will be interviewed by research assistant(s). Themes of qualitative questions include: (1) barriers and difficulties in the set-up of the system; and (2) the concerns in choosing wireless or cable connection for the monitoring device. Meanwhile, when the main trial ends, a total of 8-10 care staff from all participating units responsible to operate the system will be interviewed about their perceived benefits and acceptability of the system. Themes of qualitative questions include: (1) Acceptance of using the remote health monitoring system (including ease of operation, care staff's confidence and convenience in using the system); (2) Benefits of using the remote health monitoring system (including usefulness of the innovation, impacts on quality of care); (3) Concerns in using the remote health monitoring system (including if any residents stop using the sensor and the reason behind); and (4) Overall perception of using the remote health monitoring system. For both parts of the qualitative sub-study, an interview guide with open-ended and iterative questions will be used to probe for more experiences from the interviewees. Each interview will be conducted by a trained research assistant and will last about 15 - 30 minutes.

Blinding

Blinding is not applicable in this single group study.

Sample size determination

The sample size is estimated by the number and availability of the staff in the participating units. It is estimated that a total of 10-12 staff will be recruited.

Data analyses

The proportion of all the responses in the staff survey will be calculated. The number of abnormal vital signs, hospital admission and further medical assistance due to the adoption of the system will be counted.

The qualitative interview content will be transcribed verbatim in Chinese for further analysis. The qualitative interview transcripts will be analyzed using framework analysis to construct a coherent and logical structure from the classification of many opinions and perceptions of the system. The results will then be discussed and consolidated in the panel meetings with the co-authors.

ELIGIBILITY:
Inclusion Criteria for main trial:

* All care staff in Haven of Hope Woo Ping Care & Attention Home and Haven of Hope Nursing Home who are responsible to operate remote real-time health monitoring system will be invited to participate.

Inclusion Criteria for qualitative study about experience of setting up the system:

* The Unit in-charge and care staff responsible to set up the system from each of the participating units will be recruited.

Inclusion Criteria for qualitative study about the operation of the system:

* All care staff joining the main trial will be recruited.

Exclusion Criteria:

* No

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study populations are all care staff who are responsible to operate remote health monitoring system in Haven of Hope Woo Ping Care & Attention Home and Haven of Hope Nursing Home.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yee Tak Cheung, PhD, Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Haven of Hope Nursing Home, Hong Kong
  - Kai Tak Holding Centre Zone D, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Research data and documentation will be available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available for 10 years.

REFERENCES:
- [Background] Piau A, Campo E, Rumeau P, Vellas B, Nourhashemi F. Aging society and gerontechnology: a solution for an independent living? J Nutr Health Aging. 2014 Jan;18(1):97-112. doi: 10.1007/s12603-013-0356-5. PMID 24402399
- [Background] Carmeli, E. Aspects of assistive gerontechnology. Int J Disabil Hum Dev. 2009; 8(3): 215-218.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants will be recruited in the elderly residential setting and community isolation facility. The recruitment period of each test sites is one week. They also need to be able to read and understand Chinese.
Pre-assignment Details: Failure to read and understand Chinese will deter smooth communication and undermine the objectivity of the study
Groups:
- Single-group: All care staff who manage the system will complete a very brief survey (1-minute) after each work shift for 14 days. Detection of abnormal vital signs will be recorded by the system. Hospital admission and further medical assistance due to the use of the system will be documented by the care team. The staff will be interviewed about their perceived benefits and acceptability of the system.
  remote real-time health monitoring system with ring-like sensor: The remote monitoring system will constantly record the temperature, pulse and oxygen saturation (SpO2) of the residents wearing the equipment. When the staff find abnormal vital signs, they will provide further medical assistance. All care staff who manage the system will be complete a very brief survey (1-minute) after each work shift for 14 days.
Period: Overall Study
Arm/Group | Single-group
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single-group
Number analyzed (Participants) | 20
Age, Customized [Count of Participants; unit: Participants]
  Age group: <30 years | 6
  Age group: 30-39 years | 3
  Age group: 40-49 years | 2
  Age group: 50-59 years | 4
  Age group: ≥60 years | 3
  Age group: Did not report | 2
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 4
  Female | 13
  Did not report | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 20
Region of Enrollment [Number; unit: participants]
  Hong Kong | 20

OUTCOME MEASURES:

1. Primary Outcome: Average Staff Perceived Overall Time-saving of the System Over 14 Days
Description: After every shift for 14 days, the staff fill in a survey for the following item with 5-point Likert scale (5= Strongly Agree, 1= Strongly Disagree):
  3. The remote real-time health monitoring system reduces your time for measuring vital signs of the residents in the previous shift
Time Frame: every day during the 2-week trial period
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Single-group
Number analyzed (Participants) | 20
Scores on a scale | 2.8 (0.9)

2. Primary Outcome: Average Staff Perception of the System on Early Detection of Abnormal Vital Signs Over 14 Days
Description: After every shift for 14 days, the staff fill in a survey for the following item with 5-point Likert scale (5= Strongly Agree, 1= Strongly Disagree):
  2. The remote real-time health monitoring system facilitates you to monitor the vital signs in the previous shift
Time Frame: every day during the 2-week trial period
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Single-group
Number analyzed (Participants) | 20
Scores on a scale | 2.8 (0.9)

3. Primary Outcome: Average Staff Perception of the System on Its Facilitation of Early Delivery of Medical Support Over 14 Days
Description: After every shift for 14 days, the staff fill in a survey for the following item with 5-point Likert scale (5= Strongly Agree, 1= Strongly Disagree):
  1. The remote real-time health monitoring system facilitates you to provide early delivery of medical support in the previous shift
Time Frame: every day during the 2-week trial period
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Single-group
Number analyzed (Participants) | 20
Scores on a scale | 2.8 (0.8)

4. Secondary Outcome: Number of Hospital Admissions and Further Medical Assistance
Description: Number of hospital admissions and further medical assistance due to the use of the system, according to hospitalization record
Time Frame: every day during the 2-week trial period
Measure: Number; unit: events
Arm/Group | Single-group
Number analyzed (Participants) | 20
events
  Hospital admissions | 1
  Further medical assistance | 1

5. Secondary Outcome: Average Perceived Staff Stress Level Over 14 Days
Description: After every shift for 14 days, the staff fill in a survey for the following items with 5-point Likert scale (5= Strongly Agree, 1= Strongly Disagree) 4. The remote real-time health monitoring system has made you feel at ease in the previous shift (For example, you feel at ease as the system facilitates easy monitoring on the vital signs of the resident) 5. The remote real-time health monitoring system has made you feel uncomfortable in the previous shift (For example, you worry that residents might take off the sensor; bad connection or system malfunction) 6. The remote real-time health monitoring system relieves your stress in the previous shift
Time Frame: every day during the 2-week trial period
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Single-group
Number analyzed (Participants) | 20
Scores on a scale
  item 4. feel at ease | 2.8 (0.8)
  item 5. feel uncomfortable | 2.8 (0.9)
  item 6. relieves stress | 2.7 (0.8)

6. Secondary Outcome: Number of Participants Agreeing That the System Can Remote Monitor the Vital Signs of the Participants
Description: During qualitative interviews, the number of participants agreeing that the system can remote monitor the vital signs of the participants
Time Frame: at the end of 2-week trial period
Population: Interviews were conducted with 6 participants. 2 participants were invited from each of the service unit.
Measure: Count of Participants; unit: Participants
Groups:
- Staff Having Used the System: Staff who check the system for the vital signs of the participants and provide medical care when needed.
Arm/Group | Staff Having Used the System
Number analyzed (Participants) | 6
Participants
  Agreeing that the system can remote monitor the vital signs of the participants | 2
  Not agreeing that the system can remote monitor the vital signs of the participants | 4

7. Secondary Outcome: Number of Participants Agreeing That the Sensor Easily Detaches From the Participants
Description: During qualitative interviews, the number of participants agreeing that the sensor easily detaches from the participants
Time Frame: at the end of 2-week trial period
Population: Interviews were conducted with 6 participants. 2 participants were invited from each of the service unit.
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Having Used the System
Number analyzed (Participants) | 6
Participants
  Agreeing that the sensor easily detaches from the participants | 4
  Not agreeing that the sensor easily detaches from the participants | 2

8. Secondary Outcome: Number of Participants Agreeing That the Vital Signs Measured by the System Are Accurate
Description: During qualitative interviews, the number of participants agreeing that the vital signs measured by the system are accurate
Time Frame: at the end of 2-week trial period
Population: Interviews were conducted with 6 participants. 2 participants were invited from each of the service unit.
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Having Used the System
Number analyzed (Participants) | 6
Participants
  Agreeing that the vital signs measured by the system are accurate | 2
  Not agreeing that the vital signs measured by the system are accurate | 4

9. Secondary Outcome: Number of Participants Agreeing That the Size of the Sensors Fit the Participants
Description: During qualitative interviews, the number of participants agreeing that the size of the sensors fit the participants
Time Frame: at the start of 2-week trial period
Population: Interviews were conducted with 6 participants. 2 participants were invited from each of the service unit.
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Having Used the System
Number analyzed (Participants) | 6
Participants
  Agreeing that the size of the sensors fit the participants | 2
  Not agreeing that the size of the sensors fit the participants | 4

10. Secondary Outcome: Number of Participants Preferring Cable or Wireless Connection for the System
Description: During qualitative interviews, the number of participants preferring cable or wireless connection for the system
Time Frame: at the start of 2-week trial period
Population: Interviews were conducted with 6 participants. 2 participants were invited from each of the service unit.
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Having Used the System
Number analyzed (Participants) | 6
Participants
  Prefer cable connection | 6
  Prefer wireless connection | 0

ADVERSE EVENTS:
Time Frame: During the 4-week trial periods in each test site
Arm/Group | Single-group
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/40/NCT05302440/Prot_SAP_000.pdf